CLINICAL TRIAL: NCT07064395
Title: Bright Light Therapy to Reduce Sleep Disturbance and Biological Aging in Lung Cancer Patients
Brief Title: Bright Light Therapy on Sleep Health in Lung Cancer Patients
Acronym: BLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Menghua Tao, Assistant Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17849; F80046 (Other Grant/Funding Number: Henry Ford Health + Michigan State University Pilot Award)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancers
Keywords: bright light; intervention; biological age; sleep; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bright light arm (Experimental): Participants will receive a daily 30-minutes bright light through light visor for 4 weeks.
  Interventions: Other: bright light
- control arm (No Intervention): Participants will not receive bright light, and keep their usual daily light exposure for 4 weeks.

INTERVENTIONS:
Other: bright light — Lung cancer patients in the bright light arm will receive 12,000 lux bright light through light visor for 4 weeks.
  Arms: bright light arm

SUMMARY:
The goal of this randomized intervention trial is to determine the effect of bright light therapy on sleep disturbance, as well as to investigate the impacts of bright light therapy on biological age measured by clinical biomarkers. The main questions it aims to answer are:

* Does bright light therapy improve sleep patterns (i.e., sleep onset latency, sleep disturbance, and sleep efficiency) in lung cancer patients?
* Can bright light therapy slow the rate of aging measured by biological age in lung cancer patients? Researchers will compare bright light therapy group to control group to see if bright light works to reduce sleep disturbance and decelerate biological aging.

Participants will:

* Receive bright light exposure or usual light exposure every day for 4 weeks
* Get blood draw at the baseline and at 4 weeks for clinical biomarkers tests
* Complete self-reported sleep, fatigue and stress surveys at the baseline and at 4 weeks
* Keep a daily sleep log

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* Stage Ib to IIIb primary lung cancer diagnosis
* >=2 months after completion of primary therapy, patient can continue to be on maintenance/immunotherapy
* ECOG performance status is 0 or 1
* Experience problematic sleep (scores of >=8 on the Insomnia Severity Index)
* Able to understand, speak, and read English
* Sighted and mentally competent to consent

Exclusion Criteria:

* Pregnant women
* Have metastatic cancer
* on oxygen therapy
* Current diagnosis of seasonal affective disorder or substance abuse
* Engage in shift work or travel across >3 time zones within 2 weeks prior to the study
* Are currently being treated for sleep apnea, restless legs syndrome, or narcolepsy
* Take prescribed sedative hypnotics or antipsychotics
* Have eye conditions (glaucoma or retinal disease), problem triggered by bright light (e.g., migraine), or take photosensitizing medications (e.g., some porphyrin drugs, antipsychotics, antiarrhythmic agents)
* Participants with an Insomnia Severity Index <8
* Participants with cognitive impairment (sores of <3 mini-cog test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in sleep patterns at 4 weeks | from enrollment to the end of the intervention at 4 weeks
  Changes in sleep patterns will be assessed by sleep efficiency (e.g., duration of sleep in hours), sleep quality (e.g., number of sleep disturbance), and sleep onset latency (e.g., minutes of falling asleep).
Changes from baseline in the measures of biological age at 4 weeks | From enrollment to the end of intervention at 4 weeks
  Participants have a lower rate of biological aging

SECONDARY OUTCOMES:
Change from Baseline in the measure of fatigue and stress at 4 weeks | From enrollment to the end of intervention at 4 weeks
  Participants will achieve a response if they have lower level of fatigue and stress level at 4 weeks. Stress will be assessed by stress scale ranging from 0 to 40, and a higher score refers to worse stress level. Fatigue will be assessed by a fatigue score ranging from 0-40, and a higher scale means severe fatigue level.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States